CLINICAL TRIAL: NCT02000453
Title: An Open Label, Experimental Medicine Investigation of the Safety and Tolerability of 400 mg b.i.d. GSK2586184 in Patients With Moderate to Severely Active Ulcerative Colitis.
Brief Title: Safety and Tolerability Study of GSK2586184 in Patients With Moderate to Severely Active Ulcerative Colitis.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: GSK has elected to terminate development principally as a result of the statin drug-drug interaction (DDI) study.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Prof Geert D'Haens, AMC, Amsterdam (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200208; 2013-001369-18 (EudraCT Number)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Colitis, Ulcerative
Keywords: Quality of Life; Infection; GSK2586184; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative; Infections | interventions — GSK2586184

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2586184 (Experimental): A total of 15 subjects to be administered 400 mg GSK2586184 Tablet (200 mg X 2) twice daily for up to 56 days
  Interventions: Drug: GSK2586184 400mg

INTERVENTIONS:
Drug: GSK2586184 400mg — White film coated round biconvex GSK2586184 200 mg tablets, administered 2 X twice daily. Tablet containing GSK2586184A, with the following excipients: microcrystalline cellulose, lactose, hypromellose, croscarmellose sodium, magnesium stearate and titanium dioxide.

SUMMARY:
This is an open label exploratory study to investigate the safety of 400 milligram (mg ) twice a day (b.i.d.) GSK2586184 in patients with moderate to severe, active ulcerative colitis (UC). Study medication will be administered orally (as tablets), twice daily, for up to 8 weeks (56 days). Study medication will be taken with food. Each subject will have 6 out-patient visits: Screening (Day -30 to -1); Baseline and Start of treatment (Day 1); Week 2 (Day 14); Week 4 (Day 28); Week 8 (Day 56); and Follow-up (Week 12; Day 84). Visit windows for weeks 2, 4 and 8 will be + 2 days. The primary objective of this study is to assess the safety and tolerability of GSK2586184. The primary endpoints to measure safety are laboratory tests (including haematology, clinical chemistry and serum creatinine), vital signs, 12-lead electrocardiogram (ECG), physical examination, and adverse event reporting. These are standard measurements to evaluate safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Moderate to severely active UC at least 6 months prior to Screening confirmed by colonoscopy or sigmoidoscopy with video recording, and biopsy.
* A Mayo score of 6 to 12 points and endoscopy sub score of 2 to 3 at screening, despite concurrent treatment with at least 1 of the following (oral corticosteroids or any oral 5-aminosalicylic acid (ASA) or both as defined below): Oral 5-ASA at a stable dose (>=2.4grams (g)/day) for at least 4 weeks from first dose. Must remain on a stable dose until end of treatment, Stable oral corticosteroid dose (prednisone of <=20 mg/day or equivalent) for at least 14 days prior to Baseline (must remain on a stable dose until end of treatment).
* Otherwise healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as: pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea.

In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milliinternational units (MlU)/milliliter (mL) and estradiol <40 picograms (pg)/mL (<147 picomole [pmol]/liter [L]) is confirmatory). Females on hormone replacement therapy (HRT) must discontinue HRT to allow confirmation of post-menopausal status before study enrollment. For most forms of HRT, at least 2 to 4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

* Male subjects with female partners of child-bearing potential must agree to use acceptable contraception methods. This criterion must be followed during the study and for at least 2 weeks after their last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Subjects with fulminant UC, or UC limited to rectum.
* Subjects with previous colonic surgery, histological evidence of colonic dysplasia, or bowel stricture.
* Subjects who have received therapeutic enema or suppository, other than required for endoscopy, within 14 days prior to the Screening endoscopy and during the remainder of Screening Period.
* Unable to refrain from the use of the prohibited drugs before the stated time before first dose of study medication until completion of the follow-up visit.
* A live vaccination within 4 weeks before the first dose of study medication, or a live vaccination planned during the course of the study (until completion of the follow-up visit).
* A major organ transplant (e.g. heart, lung, kidney, liver) or haematopoietic stem cell/marrow transplant.
* Significant unstable or uncontrolled acute or chronic disease unrelated to UC (i.e. cardiovascular including uncontrolled hypertension, hypercholesterolemia, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk.
* A planned surgical procedure that, in the opinion of the investigator, makes the subject unsuitable for the study.
* A history of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* Acute or chronic infections, as follows: Known previous, active or latent infection with Mycobacterium Tuberculosis, Currently on any suppressive therapy for a chronic infection (such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria), Hospitalisation for treatment of infection within 60 days before first dose, Use of parenteral (IV or intramuscular) antibiotics (antibacterials, antivirals, antifungals, or antiparasitic agents) within 60 days before first dose, Serologic evidence of Hepatitis B (HB) infection based on the results of testing for HBsAg, anti-HBc antibody as follows: subjects positive for HBsAg are excluded; and subjects positive for anti-HBc antibody (regardless of anti-HBs antibody status) are excluded, Positive test for Hepatitis C antibody confirmed on the same sample with a Hepatitis C third generation immunoassay or PCR. Subjects who are positive for Hepatitis C antibody, but negative when the Hepatitis C third generation immunoassay or PCR is performed on the same sample, will be eligible to participate, Subjects who are positive for Hepatitis C antibody and have a positive or indeterminate result when the Hepatitis C third generation immunoassay or PCR is performed on the same sample, will not be eligible to participate.
* A positive test for HIV antibody.
* Haemoglobin <11 g/decilitre (dL) (6.83 millimoles[mmol]/L), haematocrit <30%, white blood cells (WBC) count (absolute) <3×10^9/L, neutrophils <1.5×10^9/L, platelets <100×10^9/L, lymphocytes<1×10^9/L.
* Current or history of renal disease, or estimated creatinine clearance <60 mL/min/1.73m^2 or serum creatinine >1.5 upper limit of normal (ULN).
* Single QT duration corrected (QTc) >450 millisecond (msec); or QTc >480 msec in subjects with Bundle Branch Block.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Alanine aminotransferase (ALT) >2xULN; alkaline phosphatase and bilirubin ≥ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >168g for males or >112 g for females (8 g of alcohol is equivalent to 240mL of beer, 125mL of wine or 25mL spirits).
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer). Or if the subject plans to take part in another clinical trial at the same time as participating in this clinical trial.
* History of sensitivity to any components of the study medications, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates their participation.
* Where donation of blood or blood products, in addition to those required for the study, would be in excess of 500 mL within a 56 day period.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the consumption of grapefruit or grapefruit juice from 3 weeks before the first dose of study medication until 2 weeks after the last dose of study medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2014-08-08 (Actual); Study Completion 2014-08-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of twice daily doses of GSK2586184 | Up to Week 8
  Safety and tolerability, as determined by laboratory tests (including haematology, clinical chemistry and serum creatinine) vital signs, 12-lead Electrocardiogram (ECG), physical examination, and adverse event reporting.
Safety as assessed by the collection of adverse events (AEs) | Up to Week 8
  AEs will be collected from the start of Study Treatment and until 5 days post last-dose (at follow up).
Safety as assessed by laboratory parameters | Up to Week 8
  Laboratory parameters include hematology, clinical chemistry, urinalysis Absolute values and changes over time of hematology, clinical chemistry, urinalysis will be assessed.
Safety as assessed by vital sign measurement | Up to Week 8
  Vital signs include systolic blood pressure, diastolic blood pressure, temperature, and heart rate.
Safety as assessed by ECG rhythm. | Up to Week 8
  Continuous monitoring of a subject' heart rate and rhythm by ECG.

SECONDARY OUTCOMES:
Efficacy of GSK2586184 in achieving clinical and endoscopic remission after 8 weeks of treatment | Up to Week 8
  Efficacy assessed by total Mayo score of 2 points or lower, with no individual sub score exceeding 1 point, and reduction in endoscopic mucosal appearance score of >= 1.
Efficacy of GSK2586184 in achieving symptomatic clinical remission after 8 weeks | Up to Week 8
  Efficacy assessed by Mayo score for the proportion of subjects who achieve a score of 0 for both rectal bleeding and stool frequency.
Efficacy of GSK2586184 in achieving clinical response | Up to Week 8
  Efficacy assessed by Mayo score for the proportion of subjects of subjects who achieve a decrease from baseline in total Mayo score of >=3 points, with an accompanying decrease in the sub score for rectal bleeding of at least 1 point or an absolute sub score for rectal bleeding
Efficacy of GSK2586184 in achieving mucosal healing. | Up to Week 8
  Efficacy assessed by proportion of subjects who achieve an absolute sub score for endoscopy of 0 or 1, at week 8. And change from baseline of mucosal appearance determined by ulcerative colitis endoscopic index of severity (UCEIS).
The effect of twice daily doses of GSK2586184 on health related quality of life (QoL) in UC patients. | Up to Week 8
  Change from baseline of inflammatory bowel disease questionnaire (IBDQ) was assessed
The effect of twice daily doses of GSK2586184 on serum C reactive protein (CRP) levels in UC patients | Up to Week 8
  Change from baseline in mean serum CRP levels was assessed.
The effect of twice daily doses of GSK2586184 on faecal calprotectin levels | Up to Week 8
  Change from baseline of mean faecal calprotectin levels was assessed.
The plasma pharmacokinetics of repeated, twice daily doses of GSK2586184 | Up to Week 8
  Plasma concentrations and derived pharmacokinetic parameters of GSK2586184 were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Amsterdam, Netherlands

REFERENCES:
- [Background] De Vries LCS, Ludbrook VJ, Hicks KJ, D'Haens GR. GSK2586184, a JAK1 selective inhibitor, in two patients with ulcerative colitis. BMJ Case Rep. 2017 Aug 7;2017:bcr2017221078. doi: 10.1136/bcr-2017-221078. PMID 28790099